CLINICAL TRIAL: NCT04770558
Title: Effectiveness of Interactive Exergame to Improve Physical and Cognitive Functions in Older Adults With Sarcopenia
Brief Title: Effectiveness of Interactive Exergame in Older Adults With Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Shu-Chun Lee, Assistant Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N202012029
Record Dates: First submitted 2021-02-21; First posted 2021-02-25 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame group (Experimental): The exergame group will receive exergame training for 12 weeks, 2 times a week and 60 min per session.
  Interventions: Other: Interactive Exergame
- Control group (No Intervention): The control group will not receive any intervention and maintain their lifestyle for 12 weeks.

INTERVENTIONS:
Other: Interactive Exergame — The one-to-one supervised training session consists of 10 min warm-up exercise, 40 min interactive exergame, and 10 min cool-down exercise. Both physical (muscle strength, coordination and balance in lower limbs) and cognitive functions (visuospatial, attention, short-term memory, calculation, reaction and executive function) will be trained through the interactive exergame.
  Arms: Exergame group

SUMMARY:
Sarcopenia has been defined as an age related, involuntary loss of skeletal muscle mass and strength. The prevalence of sarcopenia is about 10% globally, and risk factors of sarcopenia includes age, lower physical activity, and malnutrition. Sarcopenia can lead to many adverse health outcomes, particularly in physical and cognitive functions. Most of previous studies have reported that interactive exergame can improve cognitive and physical functions in older population but none of studies use of interactive exergame on older adults with sarcopenia. Therefore, the aim of study will investigate the effects of interactive exergame on older adults with sarcopenia.

DETAILED DESCRIPTION:
A total of 60 older participants will be randomly assigned to the experimental and control groups. Participants in the experimental group will receive 40 minutes per session, 2 times a week for 12 weeks interactive exergame while those in the control group will maintain their regular activity. All participants will be assessed their physical and cognitive function, sarcopenia index and other health related outcome measurements before and after intervention program.

ELIGIBILITY:
Inclusion Criteria:

1. 65-99 years old
2. able to walk 6 meters without assistance devices
3. older adults with possible sarcopenia, sarcopenia or severe sarcopenia

Exclusion Criteria:

1. people with hemodialysis
2. people with built-in electronic medical equipment
3. people with central nervous system disease such as stroke or Parkinson's disease
4. score in ascertain dementia 8 more than 2
5. people with mental illness

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-01-11 (Estimated); Study Completion 2022-01-11 (Estimated)

PRIMARY OUTCOMES:
Hand grip | Change from Baseline hand grip at Week 12
  Dominant hand grip (kg) will measured by a dynamometer. Participants will stand with their arms down by their sides. They will squeeze the dynamometer with maximum isometric effort, which is maintained for 6 seconds.
  Female less than 18 kg and man less than 28 kg indicate weakness in grip strength.
Lower limbs strength | Change from Baseline lower limbs strength at Week 12
  Lower limbs strength will be assessed by the Five Times Sit to Stand. Participants will be asked to sit on the chair with arms folded across their chest, and stand up and sit down as quickly as possible for 5 times. The time (s) to complete the task will be recorded.The time more than 12 seconds indicates weakness in lower limbs strength.
Appendicular muscle mass | Change from Baseline appendicular muscle mass at Week 12
  Appendicular muscle mass will be assessed by the Body Impedance Analysis (BIA).Participants will be asked to stand on the machine and hold the handle of the machine. Female less than 5.7kg/m2 and male less than 7 kg/m2 indicate lower muscle mass.
Function ability | Change from Baseline function ability at Week 12
  Function ability test will be determined by the timed up and go test (TUG). Participants will be asked to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. The times(s) to complete the task will be recorded. Higher than 12s indicate weakness in function ability.
Static balance | Change from Baseline static balance at Week 12
  Static balance test will be assessed by the modified Clinical Test for Sensory Interaction in Balance(mCTSIB), The mCTSIB was developed as a clinical version of the Sensory Organization Test and was developed to assesses sensory contributions to postural control.
  Participants will stand with their hands at their sides, feet together and perform the following 4 sensory conditions: (1) Stand on firm surface with eyes open (2) Stand on firm surface with eyes closed (3) Stand on foam surface with eyes open (4) Stand on foam surface with eyes closed. Each condition will be timed for maximum 30 seconds. The test is terminated when a participant's arms or feet moves. If participants are unable to maintain the position for 30 seconds, they are then provided with 2 additional attempts. The time (s) to complete each condition will be recorded.If they can't complete this test indicate weakness in static balance
Walking ability | Change from Baseline walking ability at Week 12
  Walking ability test will be measured by the 6 meter walk test. Participant will be asked to walk at their self-selected speed. The time for the middle 6 meters will be recorded and walking speed (m/s) will be calculated.
Fear of falling | Change from Baseline fear of falling at Week 12
  Fear of falling will be measured by the Falls Efficacy Scale- International (FES-I). The FES-I rates each daily task from "no confident at all" to "completely confident". The total score is between 16 and 64, and the score more than 28 indicates higher level of fear of falling.
Cognitive function | Change from Baseline cognitive function at Week 12
  Cognitive function will be evaluated by the Montreal Cognitive Assessment (MoCA), which includes visuospatial abilities, short-term memory recall task, multiple aspects of executive functions, attention, concentration, and working memory. The total score is 30 and the score less than 26 indicates mild cognitive impairment.

SECONDARY OUTCOMES:
Physical Activity | Change from Baseline physical activity at Week 12
  Physical Activity will be examined by the International Physical Activity Questionnaire (IPAQ)-Short Form. Participants will be asked about their duration (in minutes) and frequency (days) when performing four specific types of activity: walking, moderate intensity, vigorous intensity and sitting. Female less than 270 kcal and male less than 383 kcal indicate low physical activity.
Diet record | Change from Baseline diet record at Week 12
  Diet record will be examined by the Three Day Diet Record. Participants will be asked to record their three random days' protein diet during a week, every week when they start the intervention, researchers will record their new data.
Depression | Change from Baseline depression at Week 12
  Depression will be evaluated by the Geriatric Depression Scale (GDS) consisting of 15 questions. Participants will be asked to recall their feelings about some things in the past week. The answer is "Yes" or "No". The score is calculated according to the nature of the question, and the total score is 15 points. The higher the score, the higher the degree of depression. When the score is greater than 5 points, it indicates the presence of depression.
Health-related quality of life | Change from Baseline health-related quality of life at Week 12
  Quality of life will be evaluated by the WHOQOL-BREF Taiwan version consisting of 28 questions, which is simplified from the WHOQOL long form. Two of these questions are self-evaluated quality of life and health status, other 26 questions fall into four categories (physiological, psychological, social, and environmental quality of life).The higher score and the better quality of life.

OTHER OUTCOMES:
Sarcopenia screening | Baseline
  Sarcopenia will be screened by the SARC-F questionnaire including strength, assistant in walking, rise from a chair, climb stair and fall. The answer is not difficult with 0 point, a little difficult with 1 point and very difficult with 2 points.The score is total score is between 0 and 10. The score more than 4 indicates high risk of sarcopenia.
Dementia screening | Baseline
  Dementia will be screened by Ascertain dementia 8(AD-8) including 1.problems with judgment 2.decreased interest 3.repeats 4.learning 5.forgets month or year 6.handling financial 7.trouble remembering appointments 8.problems with memory.They consider the changes in the past and the present, instead of responding to their current performance.The score more than 2 indicates high risk of dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chun Lee, PhD, Principal Investigator — School of Gerontology Health Management
Locations (1):
- Community daycare center, Taipei, Taiwan